CLINICAL TRIAL: NCT06194838
Title: Clinical Outcomes Associated With At Home Use of Non-Powered vs. Powered Prosthetic Knees by K2-level Individuals With Transfemoral Amputations
Brief Title: Clinical Outcomes With Non-Powered vs. Powered Prosthetic Knees by K2-level Amputees
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liberating Technologies, Inc. (Industry)
Collaborators: Hanger Clinic: Prosthetics & Orthotics (Other)
Responsible Party: Principal Investigator, Jennifer Johansson, Principal Investigator, Liberating Technologies, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 10877
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Amputation; Amputation; Traumatic, Leg, Lower; Limb; Absence, Congenital, Lower; Prosthesis User; Lower Limb Amputation Above Knee (Injury); Amputation; Traumatic, Leg: Thigh, Between Hip and Knee
Keywords: amputee; lower limb amputee; transfemoral amputee; prosthetic knee; power knee; mechanical knee; lower limb prosthesis user
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants will take home three interventional devices for data collection and feedback. One of the interventions will be the commercially available Ossur OFM-2, a passive mechanical knee, and the most commonly used knee for K2 users. The two other interventional devices will be commercially available powered knees: (1) the Ossur Power Knee and (2) the Reboocon Intuy Knee. Participants will be trained on the interventional knees during the first month of at-home use. Functional outcome measures and self-report surveys will also be completed in-lab before and after each take-home intervention, as well as at the last training visit, in order to form a detailed comparison between the three interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Comparator Baseline (No Intervention): The subject will wear the Ossur OFM-2, a passive mechanical knee which is the most commonly used knee for K2 users, for 3 months, as well as in the lab to complete outcome measures.
- Ossur Power Knee (Experimental): The subject will wear the Ossur Power Knee for 3 months, as well as in the lab to complete outcome measures.
  Interventions: Device: Ossur Power Knee
- Reboocon Intuy Knee (Experimental): The subject will wear the Reboocon Intuy Knee for 3 months, as well as in the lab to complete outcome measures.
  Interventions: Device: Reboocon Intuy Knee

INTERVENTIONS:
Device: Ossur Power Knee — Newest version of the commercially-available powered knee developed by Ossur.
  Other Names: Ossur Power Knee III; PK3
  Arms: Ossur Power Knee
Device: Reboocon Intuy Knee — Commercially-available powered knee developed by Reboocon.
  Other Names: Intuy Knee
  Arms: Reboocon Intuy Knee

SUMMARY:
The goal of this proposed project is to gather community-based data from the K2-level Transfemoral Amputee (TFA) population to aid in evidence-based prescription of powered prosthetic knees (i.e., choosing the right device to maximize the benefit for each patient). The investigators intend to use this trial data along with a concurrent study being conducted within the K3-K4 level population to guide the implementation of effective prescriptions towards those that can benefit most from a given device and limit prescription to those who would not see benefit in order to ensure the most judicious use of Department of Defense (DoD) and Veteran's Affairs healthcare dollars. The findings will also be shared with the research community to help drive the design of future devices by identifying what features and functions are most beneficial to which patient populations when the devices are used outside of the laboratory. In summary, more community-based data on how powered prosthetic knees compare with the current standard in TFA populations is needed to allow for improved clinical decision making and clinical outcomes.

DETAILED DESCRIPTION:
This study will focus on investigating the tradeoffs between powered knees and mechanical knees to identify the prosthetic knee that is best suited for K2 users during different tasks. The investigators will assess measured, observed, and self-reported outcomes achieved through real-world use of these prosthetic knees.

The results of this study will (1) provide initial evidence to guide clinical prescription and use of powered knee technologies for K2-level individuals with sound scientific data, (2) provide pilot data for a larger clinical trial to further inform the evidence-based prescription of powered knee technologies to other K-levels, and (3) obtain data that can be disseminated to other researchers and inform the design of future powered prosthetic knees by understanding the needs of users and identifying the features and functions that are most valuable to this patient population, as well as evaluating the capabilities and limitations of current devices.

The investigators plan to perform a pilot longitudinal randomized crossover study to compare the effects of power at the knee in individuals with unilateral transfemoral amputation. The three interventions, or conditions, to be tested are: (A) the Össur Power Knee, a powered knee that has recently released its third version, (B) The Reboocon Intuy Knee, a newly commercialized powered knee, and (C) the Össur OFM-2, a passive mechanical knee, and the most commonly used knee for K2 users. The two powered knees being tested differ in aspects such as max power/torque, weight, algorithm, and battery life. Therefore, this study will not only provide insights to the role powered knees play in the K2 population, but also if certain aspects of each powered knee are more preferred or accepted by patients in order to inform future powered knee developments and clinical treatment.

The order of the knee conditions will be randomized across subjects. Block randomization using a previously developed custom program based on random number generation will be used to equally distribute the subjects into the 6 possible intervention orders (ABC, ACB, BAC, BCA, CAB, CBA). For each condition, the subject will be trained on and acclimated to the device during the first month of the take-home period, and then will continue to wear it at home for two more months for a total of three months per condition. There may be seasonal effects due to the timing of when the various test conditions are administered, however, the investigators plan to offset these effects with condition randomization, multiple site testing, and staggered start times.

Testing will consist of test sessions, training sessions, at-home wear of the device, and functional and self-report assessment for each intervention condition.

After receiving IRB approval, subjects will be recruited and screened for eligibility. If they are eligible and decide to participate, they will be scheduled for their first site visit. They will either be consented over the phone before their first site visit or at the first site visit. If over the phone, study staff will use the telephone script to confirm eligibility and guide the subject through consent form details. Subjects will be given the informed consent form to read through entirely before signing and are encouraged to ask questions at any time.

Each subject will be provided with a standardized commercially available prosthetic ankle/foot appropriate for K2-ambulators (e.g., Össur Pro-Flex LP), to wear throughout all study periods for comparability between subjects and conditions.

Prior to each condition, each subject will be fit and aligned on the knee by a trained certified prosthetist. An activity monitor (such as the GeneActiv™) will be worn by the subject. As the investigators have done in prior studies, they will use the activity monitor to track the number of steps the subjects take during each condition.

The subject will wear the knee being tested at home for three months. During the first month of each condition, subjects will acclimate to the knee and participate in at least four, but up to eight, 1-hour training sessions. At a minimum, each subject will receive three training sessions to learn how to properly use each device for a variety of daily activities and a fourth session to demonstrate retention of the learned skills. Subjects will continue training until they show retention of the understanding and/or proficiency of the device functions or until they have received eight training sessions, whichever comes first. After eight training sessions, they will have completed all of the available training and will therefore continue with the study at their current proficiency level. Functional tests and self-report surveys will be administered at the first and last training sessions to evaluate changes in these metrics caused by the training. For each condition, the investigators will work with trained and experienced clinicians, and prosthetic knee manufacturers as needed, to develop the training protocol and determine proficiency. At the last training session, the subject will complete a subset of the outcomes and self-report measures in order to collect and compare data from before and after the subject gets trained on each knee condition.

Subjects will be asked to continue to wear the knee full time for the remainder of the three-month take-home period. The investigators will call the patient periodically to ask them whether they have experienced a recent fall. If they respond positively that they had a fall, follow-up questions may be asked via a standardized fall questionnaire similar to those used in prior studies to get more specific details. After three months of at-home wear, the subject will return for the second test visit. During that visit, functional tests and self-report surveys will be administered on the first knee. Afterwards, the fitting, training, at home wear, and in-clinic assessments described above will be repeated for the second and third knee conditions.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years old
* Transfemoral prosthesis user (limb absence between the knee and hip)
* Current user of a mechanical knee
* Regularly wears prosthesis at least 5 days per week
* Have adequate clearance between distal end and ground for necessary knee and foot components
* Current Medicare Functional Classification Level (K-Level) of 2 as determined by the healthcare team
* Socket-Comfort Score: 6 or above to ensure adequate socket fit
* Six months or more experience on a prosthesis
* Body weight between 50kg and 116kg (110lbs - 256lbs)
* Height between 1.2m and 1.95m (47.2in and 76.8in)
* Has a phone to answer periodic study calls

Exclusion Criteria:

* Present injuries to residual limb or contralateral leg affecting functional ability
* Contralateral amputation proximal to MTP (metatarsophalangeal) joint
* Socket issues/changes in the last 6 weeks
* Users with bone-anchored implants
* Health or medical condition, diagnosis, or other cause that would prevent participant from effectively following study protocol, performing required outcome measures, and/or completing the study

Subjects can be excluded at the discretion of the investigator for other unforeseen disqualifying criteria (such as specific cognitive issues, etc.).

If subjects experience a health or medical condition that leaves them immobile for more than 2 weeks, they may be given the option to restart the study condition upon recovery, as long as eligibility criteria is still met, and comparable baseline functionality is demonstrated with outcomes measures.

Using a knee that the subject is unfamiliar with may increase the risk of falling. Therefore, pregnant women should not participate in the study and will be screened by self-disclosure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Step count | Monitored over entire study (9 months)
  Prior to each condition, each subject will be fit and aligned on the designated knee by a trained certified prosthetist. An activity monitor (such as the GeneActiv™) will be worn by the subject during each 3 month intervention period. Similar to prior studies, the investigators will use the activity monitor to track the number of steps the subjects take in each condition. A higher step count is a better outcome.
Activities-Specific Balance Confidence scale (ABC) - Measuring change from baseline | Throughout study completion, an average of 9 months
  The ABC is a structured questionnaire that measures an individual's confidence during ambulatory activities without falling or experiencing a sense of unsteadiness. It consists of 16 questions gauging the individual's confidence while doing activities, from 0 (no confidence) to 4 (complete confidence). A higher score means a better outcome.
  This survey will be given at the beginning and end of each study condition (3 conditions, 3 months per condition). Additionally, this survey will be given at the subject's last training session, which is dependent on the subject's scheduling availability and proficiency with each knee condition. The subject will have between 4-8 training sessions per condition until deemed proficient or the 8th session has been completed, whichever comes first. All training sessions are expected to be completed within the first month of each condition. This survey will be administered as a part of the master questionnaire.
Prosthesis Evaluation Questionnaire - Well Being (PEQ-WB) - Measuring change from baseline | Throughout study completion, an average of 9 months
  The version of the PEQ which will be administered consists of 2 questions in 1 category (well being). For purposes of easier administration, the investigators have adopted the modified 10-point ordinal scale version of the PEQ-WB (scale 1-10, where a higher score is a better outcome).
  This survey will be given at the beginning and end of each study condition (3 conditions, 3 months per condition). Additionally, this survey will be given at the subject's last training session, which is dependent on the subject's scheduling availability and proficiency with each knee condition. The subject will have between 4-8 training sessions per condition until deemed proficient or the 8th session has been completed, whichever comes first. All training sessions are expected to be completed within the first month of each condition. This survey will be administered as a part of the master questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Johansson, MS, Principal Investigator — Liberating Technologies, Inc.
Locations (1):
- Hanger Clinic, Austin, Texas, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT06194838/ICF_000.pdf